CLINICAL TRIAL: NCT00003938
Title: A Strategic Study to Determine the Optimal Moment to Initiate Systemic Antifungal Therapy With Ambisome in Granulocytopenic Cancer Patients With Unexplained Fever Refractory to Empirical Antibacterials
Brief Title: Liposomal Amphotericin B in Treating Granulocytopenia and Persistent Unexplained Fever in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: EORTC-19951; EORTC-19951
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Cancer
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV breast cancer; stage IIIA breast cancer; monoclonal gammopathy of undetermined significance; stage IIIB breast cancer; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; recurrent childhood rhabdomyosarcoma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; stage 0 chronic lymphocytic leukemia; Waldenstrom macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; small intestine lymphoma; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; unspecified childhood solid tumor, protocol specific; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; polycythemia vera; primary myelofibrosis; essential thrombocythemia; fever, sweats, and hot flashes; childhood acute promyelocytic leukemia (M3); testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; recurrent ovarian germ cell tumor; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; ovarian yolk sac tumor; ovarian embryonal carcinoma; ovarian polyembryoma; ovarian choriocarcinoma; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; ovarian mixed germ cell tumor; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; de novo myelodysplastic syndromes; high risk metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; primary central nervous system non-Hodgkin lymphoma; neutropenia; infection; previously untreated childhood rhabdomyosarcoma; prolymphocytic leukemia; primary systemic amyloidosis; intraocular lymphoma; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; previously treated childhood rhabdomyosarcoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Hodgkin Disease; Breast Neoplasms; Monoclonal Gammopathy of Undetermined Significance; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Multiple Myeloma; Carcinoma, Ovarian Epithelial; Neuroblastoma; Wilms Tumor; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Testicular Neoplasms; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Fever; Hot Flashes; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Seminoma; Carcinoma, Embryonal; Leukemia, Hairy Cell; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Neutropenia; Infections; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Intraocular Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Lymphoma, B-Cell, Marginal Zone | interventions — liposomal amphotericin B

INTERVENTIONS:
Drug: liposomal amphotericin B

SUMMARY:
RATIONALE: Liposomal amphotericin B may be effective in controlling fever and granulocytopenia. It is not yet known which regimen of liposomal amphotericin B is more effective in treating cancer patients who have these conditions.

PURPOSE: Randomized phase III trial to compare the effectiveness of two regimens of liposomal amphotericin B in treating granulocytopenia and fever in cancer patients.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy and side effects of amphotericin B-liposomal formulation initiated 72-84 hours vs 144-156 hours after onset of a febrile episode in cancer patients with granulocytopenia and persistent unexplained fever refractory to antibacterials.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to antifungal prophylaxis (yes vs no) and type of underlying condition. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive amphotericin B-liposomal formulation IV over 1 hour on day 3 of febrile neutropenia.
* Arm II: Patients receive amphotericin B-liposomal formulation IV over 1 hour on day 6 of febrile neutropenia.

Treatment continues until signs and symptoms of the fungal infection appear or febrile neutropenia has resolved. Persistently neutropenic patients receive treatment for at least 10 days or until another cause of infection is determined.

Patients are followed weekly for 3 weeks.

PROJECTED ACCRUAL: A total of 450 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Hematologic malignancy or solid tumor
* Must be undergoing remission induction and/or consolidation therapy for hematologic malignancy only OR
* Must be undergoing allogeneic or autologous bone marrow transplantation
* Granulocyte count less than 500/mm^3 and profound granulocytopenia expected to last for greater than 5 days
* Fever (greater than 38.5 degrees C) refractory for greater than 72 hours and less than 84 hours to broad spectrum antimicrobials, after exclusion of current bacterial, fungal, viral, parasitic, and mycobacterial infections
* Peripheral blood cultures and central venous catheter cultures negative for infections
* No microbiological documentation of a bacterial infection (e.g., abscess at catheter site)
* No invasive fungal infection
* No probable noninfectious cause of fever

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Karnofsky 40-100% OR
* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No prior anaphylactic reaction to amphotericin B
* No psychological, familial, sociological, or geographical conditions that would prevent compliance
* Not pregnant or nursing
* Normal chest X-ray or normal high resolution CT scan of the lungs

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent active systemic antifungal agents or antifungal prophylaxis (e.g., azoles or polyenes)
* No prior IV amphotericin B during same neutropenic episode
* No change in antibacterial regimen within 48 hours prior to study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 1999-06; Primary Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P. Ljungman, MD, Study Chair — Karolinska Institutet
Locations (24):
- Belgium (5):
  - A.Z. St. Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - U.Z. Gasthuisberg, Leuven
  - Clinique Universitaire De Mont-Godinne, Mont-Godinne Yvoir
- University Hospital - Olomouc, Olomouc, Czechia
- France (3):
  - CHU de Caen, Caen
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Saint-Louis, Paris
- Germany (2):
  - Universitaetsklinikum Charite, Berlin
  - Virchow Klinikum Humboldt Universitaet Berlin, Berlin
- Greece (2):
  - Athens University-Laikon General Hospital, Athens
  - Hippokration Hospital, Thessaloniki
- Szent Laszlo Korhaz, Budapest, Hungary
- Hadassah University Hospital, Jerusalem, Israel
- Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova), Italy
- University Medical Center Nijmegen, Nijmegen, Netherlands
- Hospital De Santo Antonio Dos Capuchos, Lisbon (Lisboa), Portugal
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Spain (2):
  - Hospital de la Santa Cruz I Sant Pau, Barcelona
  - Hospital Central de Asturias, Oviedo
- Huddinge University Hospital, Stockholm, Sweden
- Section of Infectious Diseases, Ankara, Turkey (Türkiye)
- Tawam Hospital, Abu Dhabi, United Arab Emirates